CLINICAL TRIAL: NCT00226746
Title: A Multicenter Phase II Trial of Weekly Gemcitabine, Paclitaxel, and Hyperfractionated External Irradiation (63.80 GY) for Locally Advanced Pancreatic Cancer
Brief Title: Efficacy Study of Gemcitabine, Paclitaxel, and Irradiation in the Treatment of Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Hani Ashamalla, MD, MD, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYM # 179; AM-05
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Pancreatic Cancer; Hyperfractionated Radiation Therapy; Gemcitabine; Paclitaxel; Carcinoma, Pancreatic Ductal
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms | interventions — Paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Radiation Therapy: 63.80 Gy (1.1 Gy BID X 58 fractions), Paclitaxel: 60 mg/m2 / week by 1- hour IV infusion on days 1, 8, 15, 22, 29, and 36.
  Gemcitabine: 75 mg/m2 / week on days 1, 8, 15, 22, 29, and 36.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel and Gemcitabine (Experimental): Radiation Therapy: 63.80 Gy (1.1 Gy twice a day X 58 fractions), Paclitaxel: 60 mg/m2 / week by 1- hour IV infusion on days 1, 8, 15, 22, 29, and 36.
  Gemcitabine: 75 mg/m2 / week on days 1, 8, 15, 22, 29, and 36.
  Interventions: Drug: Paclitaxel and gemcitabine

INTERVENTIONS:
Drug: Paclitaxel and gemcitabine — Radiation Therapy: 63.80 Gy (1.1 Gy twice a day X 58 fractions) Paclitaxel: 60 mg/m2 / week by 1- hour IV infusion on days 1, 8, 15, 22, 29, and 36.
  Gemcitabine: 75 mg/m2 / week on days 1, 8, 15, 22, 29, and 36.

SUMMARY:
The purpose of this study is to find out what effects, good and bad, the chemotherapy drugs gemcitabine (Gemzar) and paclitaxel (Taxol) have in combination with twice daily radiation treatment on locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Based on our previous experience with the use of a weekly paclitaxel dose of 60 mg/m2 and hyperfractionated radiation therapy 63.8 Gy, we are conducting this study incorporating the use of Gemcitabine at a dose level of 75 mg/m2/week in addition to our prior protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed adenocarcinoma of the pancreas.
2. Patients must have locally advanced/unresectable disease based on institutional standardized criteria of unresectability.
3. Patients with residual disease after resection (R-1 or -2, micro and macroscopic residual) are eligible.
4. Patients with biliary or gastroduodenal obstruction must have drainage prior to starting chemoradiation.
5. All malignant disease must be encompassed within a single irradiation field (12 x 12 cm maximum).
6. All patients must have radiographically assessable disease.
7. Electrocardiogram (EKG), chest x-ray, abdominal computed tomography (CT)/magnetic resonance imaging (MRI) scan must be obtained within four weeks of study entry.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
9. Required entry laboratory parameters: granulocytes >/= 1,800/µl, platelet count >/= 100,000/µl, bilirubin < 2.0 mg/dL, alanine aminotransferase (ALT) < 3 x upper limit of normal, and creatinine < 3.0 mg/dL.
10. Signed study-specific consent form prior to study entry.

Exclusion Criteria:

1. Patients who have evidence of metastatic disease in the major viscera and/or peritoneal seeding or ascites.
2. Previous irradiation to the planned field; or previous chemotherapy for pancreatic cancer (Gemzar® or Taxol®).
3. Malignancy (within the past two years) except for non-melanomatous skin cancer or carcinoma in situ of the cervix, uterus, or bladder.
4. Patients who have significant infection or other coexistent medical condition that would preclude protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
One-year overall survival rate | Up to June 2010
  Follow up for survival will be done to know this outcome

SECONDARY OUTCOMES:
Occurrence of grade 3 or higher toxicity in the gastrointestinal or pulmonary | year 2010
  Follow up for occurrence of adverse events will be done to know this outcome
Occurrence of pathological response or shrinkage of the tumor (becomes resectable) | year 2010
  Follow up for tumor response will be done to know this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Hani Ashamalla, MD, FCCP, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

REFERENCES:
- [Background] Ashamalla H, Zaki B, Mokhtar B, Colella F, Selim H, Krishnamurthy M, Ross P. Hyperfractionated radiotherapy and paclitaxel for locally advanced/unresectable pancreatic cancer. Int J Radiat Oncol Biol Phys. 2003 Mar 1;55(3):679-87. doi: 10.1016/s0360-3016(02)03791-4. PMID 12573755